CLINICAL TRIAL: NCT04887740
Title: Osteoarticular Infections on Material in Children Under 16 Years Old at the CHU of Montpellier From 2014 to 2021
Brief Title: Osteoarticular Infections on Material in Children
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0183
Record Dates: First submitted 2021-05-04; First posted 2021-05-14 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Osteoarticular Tuberculoses
Keywords: Children
MeSH Terms: conditions — Tuberculosis, Osteoarticular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The management of osteoarticular infections on equipment is complex. In order to optimize the management of these infections, the French National Authority for Health (HAS) has published good practice recommendations for prosthesis infections in adults. However, in the pediatric population, this type of infection is rarer and their management less well codified.

The aim of this retrospective and descriptive monocentric study is to identify all osteoarticular infections in children under 16 years of age managed at the Montpellier University Hospital from 2014 to 2021, to study the epidemiology and bacterial ecology of these infections and to evaluate the effectiveness of the therapeutic strategy and side effects, long-term sequels

ELIGIBILITY:
Inclusion criteria:

* osteoarticular infections on material in children under 16 years old
* hospitalized at the CHU of Montpellier

Exclusion criteria:

* over 16 years of age
* other types of osteoarticular infections

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients under 16 years old hospitalized at the CHU of Montpellier
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with incidence of osteoarticular infections | day 1
  To evaluate the incidence of osteoarticular infections on equipment in children under 16 years of age and their medical and surgical management

SECONDARY OUTCOMES:
Number of Participants with Epidemiology of osteoarticular infections | day 1
  To evaluate the Epidemiology of osteoarticular infections on material at the University Hospital of Montpellier
Number of Participants with bacterial ecology of osteoarticular infections | day 1
  To evaluate the bacterial ecology of osteoarticular infections on material at the University Hospital of Montpellier

CONTACTS AND LOCATIONS:
Overall Officials: Léa DOMITIEN, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC